CLINICAL TRIAL: NCT04588662
Title: A Prospective Natural History Study in Uveal Melanoma
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAR5976
Record Dates: First submitted 2020-07-16; First posted 2020-10-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Residual tissue samples from clinical care biopsies that would otherwise be discarded will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uveal Melanoma: Diagnosis of uveal melanoma Ability to provide written informed consent for participation in the prospective registry OR an institutional waiver by the IRB/ethics committee for retrospective data collection without written informed consent

SUMMARY:
The overall objective of this proposal is to develop and utilize a multicenter UM registry that will, in a longitudinal fashion, capture prospective data in order to characterize the natural history of UM and provide data that will be used to support the development of novel therapies for this disease. The care of patients with UM requires a multi-disciplinary team of physicians that commonly requires the involvement of both radiation oncology and interventional radiology, and is typically directed by an ophthalmologic oncologist at time of initial diagnosis of primary disease. Overall management is transitioned to a medical oncologist when distant recurrence is identified. In the case that a patient presents with metastasis at the time of diagnosis, a medical oncologist typically directs overall management. The management of surveillance for the development of metastasis following the treatment of primary disease is variable and, if performed at all, is managed by either an ophthalmologic oncologist or medical oncologist. Thus, the successful development of a registry that aims to capture the data regarding the full natural history of UM requires a collaborative effort including leaders from both the UM ophthalmologic oncology and medical oncology fields. To this end, the investigators have built an initial consortium of key ophthalmologic oncology and medical oncology leaders from multiple major UM centers in the United States.

DETAILED DESCRIPTION:
Uveal melanoma (UM) is the most common primary intraocular malignancy in adults, accounting for 85% to 95% of ocular melanoma cases. However, UM represents only about 3% to 5% of all melanomas in the United States (US). UM most commonly arises from choroidal melanocytes (85-90%), but can also arise from the iris (3-5%) and ciliary body (5-8%). The median age of diagnosis is approximately 62; however, the peak range for diagnosis is between 70 and 79. Males have a 30% greater incidence than females. A variety of putative risk factors have been identified, including the presence of light eyes, fair skin, an inability to tan, ocular melanocytosis, dysplastic nevus syndrome, and germline BRCA1-associated protein 1 (BAP1) mutations.

Importantly, there are no recent or on-going multi-center natural history studies being conducted in this disease, and this effort is the only one to be launched with the goal of capturing the complete course of this disease, from diagnosis, initial management, surveillance, and treatment of recurrent disease in a national and international setting. This registry is especially important in providing such needed data.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of uveal melanoma
* Ability to provide written informed consent for participation in the prospective registry OR an institutional waiver by the IRB/ethics committee for retrospective data collection without written informed consent

Exclusion Criteria

*None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Diagnosis of uveal melanoma
  * Male/Female over the age of 18 years of age
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Relapse-free Survival Rate | Up to Five years
  Document the relapse-free survival of patients with uveal melanoma from the time of diagnosis of primary disease
Overall Survival Rate | Up to Five years
  document the overall survival of patients with uveal melanoma from the time of diagnosis of primary disease
Overall Survival Rate of Patients with Uveal Melanoma | Up to Five years
  document the overall survival of patients with uveal melanoma from the time of development of metastatic disease

CONTACTS AND LOCATIONS:
Overall Officials: Mariam El-Ashmawy, MD, PhD, Principal Investigator — Columbia University
Locations (17):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Australia (8):
  - Royal Adelaide Hospital, Adelaide
  - Chatswood Eye Specialists, Chatswood
  - Royal Victorian Eve and Ear Hospital, East Melbourne
  - Western Eye Specialists, Maribyrnong
  - Pennington Eye Clinic, North Adelaide
  - Perth Retina, Subiaco
  - Dr. Conway Private Rooms, Sydney
  - St. Vincent's Hospital, Sydney
- Princess Margaret Cancer Center, Toronto, Canada
- Erlangen, Erlangen, Germany
- United Kingdom (3):
  - Clatterbridge Cancer Centre, Birkenhead
  - Mount Vernon Cancer Centre, Northwood
  - Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided